CLINICAL TRIAL: NCT05805488
Title: Evaluation of the Body Slimming Effect of Lactobacillus Delbrueckii Ssp. Bulgaricus TCI904
Brief Title: Evaluation of the Body Slimming Effect of TCI904
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CMUH110-REC2-070
Record Dates: First submitted 2023-03-27; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Body Weight; Metabolic Syndrome
MeSH Terms: conditions — Body Weight; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo sachet (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo sachet
- TCI904 sachet (Experimental)
  Interventions: Dietary Supplement: TCI904 sachet

INTERVENTIONS:
Dietary Supplement: Placebo sachet — consume 1 sachet per day
  Arms: Placebo sachet
Dietary Supplement: TCI904 sachet — consume 1 sachet per day
  Other Names: Lactobacillus delbrueckii ssp. bulgaricus TCI904
  Arms: TCI904 sachet

SUMMARY:
To assess the efficacy of Lactobacillus delbrueckii ssp. bulgaricus TCI904 on body slimming

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20
* BMI ≥ 23 or male body fat ≥ 25%, female body fat ≥ 30%.
* History of Atherosclerotic cardiovascular disease (including cerebrovascular disease, coronary heart disease, peripheral vascular disease) or Type 2 diabetes or have any of the following factors: Age Men ≥ 45 years, Women ≥ 55 years or amenorrhea, hypertension, hyperlipidemia (total cholesterol > 200 mg/dL or low-density lipoprotein cholesterol LDL-C > 130 mg/dL or triglyceride TG > 130 mg/dL), high-density lipoprotein cholesterol HDL-C < 40 mg/dL.
* If people have routinely taken drugs for lowering blood sugar, blood pressure or blood lipids, there is no significant dose change within three months (variation ≤ 20%).
* Volunteers who are willing to participate in and complete the trial plan after explaining by the researchers, and sign the consent form.

Exclusion Criteria:

* History of diabetic ketoacidosis.
* Medical records documented cerebrovascular disease, acute myocardial infarction or coronary artery bypass surgery or placement of coronary artery stents or peripheral vascular disease within the last 6 months.
* Known acute infectious illness within the past month with > 7 days of antibiotics.
* Known short-term use of steroids, NSAIDs, anti-rejection drugs, interferon, immunomodulators or changes in long-term doses due to any factors in the past month.
* Have used any weight loss drugs (including Orlistate, Lorcaserin, liraglutide) within the past three months.
* History of any cancer in the past 5 years or still receiving cancer treatment.
* Patients with abnormal liver function (GOT or GPT greater than 3 times the upper limit of normal) or known cirrhosis.
* Patients with abnormal kidney function (eGFR < 30 mL/min/1.73 m^2).
* Patients with a history of alcoholism.
* Have participated in any other interventional clinical research within the last month.
* Pregnant and lactating women.
* Known history of allergy to the test substance.
* Patients who are judged inappropriate by the trial host.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The change of body weight (kg) | Week 0, week 12
  The body weight was assessed by Body Composition Monitor
The change of BMI (kg/m^2) | Week 0, week 12
  The BMI was assessed by Body Composition Monitor
The change of body fat rate (%) | Week 0, week 12
  The body fat rate was assessed by Body Composition Monitor

SECONDARY OUTCOMES:
The change of total cholesterol | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of total cholesterol
The change of triglyceride | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of triglyceride
The change of HDL-C | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of HDL-C
The change of LDL-C | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of LDL-C
The change of blood glucose | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of glucose
The change of C-reactive protein | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of C-reactive protein
The change of insulin | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of insulin
The change of HbA1c | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of HbA1c
The change of TNF-alpha | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of TNF-alpha
The change of Hypoxia-inducible factor 1-alpha (HIF-1alpha) | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of HIF-1alpha
The change of cyclooxygenase-2 (COX-2) | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of COX-2
The change of Matrix metalloproteinase (MMP) | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of MMP
The change of aspartate aminotransferase | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of aspartate aminotransferase
The change of alanine aminotransferase | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of alanine aminotransferase
The change of albumin | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of albumin
The change of creatine | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of creatine
The change of blood urea nitrogen (BUN) | Week 0, week 12
  Fasting venous blood was sampled to measure concentrations of BUN

CONTACTS AND LOCATIONS:
Overall Officials: Yang-Chang Wu, Principal Investigator — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan